CLINICAL TRIAL: NCT02790814
Title: Evaluation of an Innovative Fetal Heart Rate Monitoring Device (Named Moyo) to Improve Perinatal Outcome at Haydom Hospital, Tanzania
Brief Title: Moyo; strap-on Fetal Heart Rate Monitoring in a Rural Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Moyo Rural
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moyo strap-on (Experimental): Continous fetal heart rate monitoring
  Interventions: Device: Moyo strap-on
- Hand-held fetoscope (Active Comparator): Intermittent fetal heart rate monitoring
  Interventions: Device: Hand-held fetoscope

INTERVENTIONS:
Device: Moyo strap-on — Continous measurements
  Arms: Moyo strap-on
Device: Hand-held fetoscope — Intermittent measurements
  Arms: Hand-held fetoscope

SUMMARY:
Annually, an estimated 2.6 million still births occur half of which die during labor and delivery (fresh stillbirths). In addition, around 750,000 newborns die shortly after birth due to intrapartum-related hypoxia or birth asphyxia. Almost 99% of these perinatal deaths take place in low-income countries where the provider/patient ratio is low and fetal monitoring is inadequate. Poor intrapartum fetal heart rate monitoring, failure to identify fetal distress, and subsequently intervene, is a common pathway to perinatal deaths in these low-resourced settings. Recently, an innovative fetal heart rate monitoring device, called Moyo, using ultrasound technology, was developed to be strapped on the mother during labour. This project will compare the effectiveness of automatic use of Moyo versus intermittent use of hand-held fetoscope in detection of abnormal fetal heart rate, through a randomized control study, at Haydom Hospital, Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Women admitted in labor

Exclusion Criteria:

* Women scheduled for elective cesarean section, women with abnormal fetal heart rate on admission, multiples, and critically ill patients with no measurements of fetal heart rate on admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2652 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Frequency of abnormal fetal heart rate detection | Up to delivery

SECONDARY OUTCOMES:
Mode of delivery: vaginal versus operative | Up to delivery
Neonatal outcome: dead versus alive | Up to 24 hours
Time from abnormal fetal heart rate detection to delivery in minutes | Up to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hege L. Ersdal, Md PhD, Study Director — Helse Stavanger HF
Locations (1):
- Haydom Lutheran Hospital, Research Institute, Haydom, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mdoe PF, Ersdal HL, Mduma E, Moshiro R, Dalen I, Perlman JM, Kidanto H. Randomized controlled trial of continuous Doppler versus intermittent fetoscope fetal heart rate monitoring in a low-resource setting. Int J Gynaecol Obstet. 2018 Dec;143(3):344-350. doi: 10.1002/ijgo.12648. Epub 2018 Sep 4. PMID 30120775